CLINICAL TRIAL: NCT04839965
Title: A Randomized, Double-Blinded, Placebo Controlled Phase II Study to Evaluate the Safety and Efficacy of IV Ampion in Adult COVID-19 Patients Requiring Oxygen Supplementation
Brief Title: Study of Intravenous Ampion in Adult COVID-19 Patients Requiring Supplemental Oxygen
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The AP-017 study was prematurely terminated by the sponsor after an interim analysis.
Sponsor: Ampio Pharmaceuticals. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP-017
Record Dates: First submitted 2021-04-08; First posted 2021-04-09 (Actual); Results first posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — aspartyl-alanyl-diketopiperazine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IV Ampion (Experimental): Ampion administered via intravenous infusion
  Interventions: Biological: Ampion
- IV placebo (Placebo Comparator): Placebo administered via intravenous infusion
  Interventions: Other: Saline

INTERVENTIONS:
Biological: Ampion — Ampion administered via intravenous infusion
  Arms: IV Ampion
Other: Saline — Placebo administered via intravenous infusion
  Arms: IV placebo

SUMMARY:
This is a Phase 2 randomized study to evaluate the safety and efficacy of IV Ampion in improving the clinical course and outcomes of adult COVID-19 patients requiring supplemental oxygen.

DETAILED DESCRIPTION:
Ampion is the low molecular weight filtrate of human serum albumin with the in vitro ability to modulate inflammatory cytokine levels. Ampion has the potential to improve clinical outcomes for COVID-19 patients by reducing inflammatory cytokines correlated with the disease.

This study aims to evaluate Ampion and clinical outcomes in patients with COVID-19 requiring supplemental oxygen.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 18 years old
2. Diagnosed with COVID-19, as evaluated by laboratory diagnostic test or diagnosis based on radiological clinical findings
3. Baseline severity categorization of severe or critical COVID-19 infection per FDA Guidance for developing drugs and biological products for COVID-19 (February 2021)

   1. Severe COVID-19

      * Symptoms suggestive of severe systemic illness with COVID-19, which include shortness of breath or respiratory distress
      * Clinical signs indicative of severe systemic illness with COVID-19, such as respiratory rate ≥ 30 per minute, heart rate ≥ 125 per minute, SpO2 ≤ 93% on room air at sea level (SpO2 ≤ 90% at altitude) or PaO2/FiO2 < 300
   2. Critical COVID-19

      * Oxygen delivered by high-flow nasal cannula (heated, humidified, oxygen delivered via reinforced cannula at flow rates >20 l/min with fraction oxygen ≥ 0.5) or
      * Non-invasive mechanical or endotracheal mechanical ventilation
4. Informed consent obtained from the patient or the patient's legal representative

Exclusion Criteria:

1. As a result of the medical review and screening investigation, the Principal Investigator considers the patient unfit for the study and/or progression to death is imminent and inevitable irrespective of the provision of treatments.
2. Clinical diagnosis of respiratory failure (therapy not able to be administered in setting of resource limitation)
3. Shock defined by systolic blood pressure <90 mm Hg, or diastolic blood pressure <60 mm Hg or requiring vasopressors.
4. Multi-organ dysfunction/failure
5. Patient has severe chronic obstructive or restrictive pulmonary disease (COPD) (as defined by prior pulmonary function tests), chronic renal failure, or significant liver abnormality (e.g., cirrhosis, transplant, etc.).
6. Patient has chronic conditions requiring chemotherapy or immunosuppressive medication.
7. A history of allergic reactions to human albumin (reaction to non-human albumin such as egg albumin is not an exclusion criterion) or ingredients in 5% human albumin (N-acetyltryptophan, sodium caprylate).
8. Prolonged QT interval.
9. Patient has known pregnancy or is currently breastfeeding.
10. Patient planning to become pregnant, or father a child, during the treatment and follow-up period and/or is not willing to remain abstinent or use contraception.
11. Participation in another clinical trial (not including treatments for COVID-19 as approved by the FDA through expanded access, emergency, or compassionate use), or participation in a trial such that enrollment in this study would fall within the time frame of the half-life of the other investigational product(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-04-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ampio Pharmaceuticals, Englewood, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- IV Ampion: Ampion administered via intravenous infusion
  Ampion: 125 mL Ampion administered via intravenous infusion twice daily (250 mL / day) for five days.
- IV Placebo: Placebo administered via intravenous infusion
  Saline: 125 mL Placebo administered via intravenous infusion twice daily (250 mL / day) for five days.
Period: Overall Study
Arm/Group | IV Ampion | IV Placebo
Started | 21 | 15
Completed | 14 | 9
Not Completed | 7 | 6
Not completed — Death | 6 | 6
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Ampion | IV Placebo | Total
Number analyzed (Participants) | 21 | 15 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (10.0) | 53.4 (15.0) | 55.4 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 14 | 13 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 20 | 12 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 18 | 14 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 15 | 36
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 37.3 (13.7) | 31.4 (6.8) | 34.9 (11.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Occurrence of Mechanical Ventilation or Death
Description: Assess the effect of Ampio compared to placebo on prevention of need for mechanical ventilation or death. This is measured as the occurrence of subjects on mechanical ventilation or death by day 28.
Time Frame: Day 28
Population: Intent to Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ampion | IV Placebo
Number analyzed (Participants) | 21 | 15
Participants | 5 | 5

2. Secondary Outcome: The Number of Participants With Treatment Emergent Adverse Events of Ampion Compared to Placebo
Description: Number of subjects with treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) of treatment of IV Ampion compared to Placebo. AEs were assessed based on symptoms as a severity rating of mild, moderate, or severe. The relationship between AE and study drug was determined as either unrelated, possibly related, or related. SAEs are defined as resulting death, life threatening, requires prolonged hospitalization, results in persistent or significant disability/incapacity, or results in congenital anomaly/birth defect.
Time Frame: Baseline to Day 60
Population: Intent to Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ampion | IV Placebo
Number analyzed (Participants) | 21 | 15
Participants
  Treatment Emergent Adverse Events (TEAE's) | 15 | 12
  Study Drug Related TEAE's | 0 | 3
  Moderate or Severe TEAE's | 12 | 8
  Serious Adverse Events | 11 | 8

ADVERSE EVENTS:
Time Frame: 60 days
Description: Patients were followed for the occurrence of Adverse Events for 60 days following the first dose of study medication.
Arm/Group | IV Ampion | IV Placebo
All-Cause Mortality (participants affected / at risk) | 6/21 | 6/15
Serious Adverse Events (participants affected / at risk) | 11/21 | 8/15
Other Adverse Events (participants affected / at risk) | 15/21 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Ampion (N=21) | IV Placebo (N=15)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 4 (4)
Cardio Respiratory Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Organ Failure (General disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Perirectal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 2 (2) | 3 (3)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Ampion (N=21) | IV Placebo (N=15)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Bandaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 5 (5) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Deafness Bilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Frequent Bowel Movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Feeling Abnormal (General disorders) | 0 (0) | 1 (1)
Feeling Hot (General disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Infusion Site Coldness (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Systemic Inflammatory Response Syndrom (General disorders) | 1 (1) | 0 (0)
Oral Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Serratia (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Tract Infection Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Infusion Related Reactions (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood Creatine Increased (Investigations) | 0 (0) | 1 (1)
Cardiac Murmur (Investigations) | 1 (1) | 0 (0)
Fibrin D Dimer Increased (Investigations) | 0 (0) | 1 (1)
Platelet Count Decreased (Investigations) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 2 (2) | 0 (0)
Weight Decreased (Investigations) | 1 (1) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Alkalosis Hypochloraemic (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Balance Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness Exertional (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Intensive Care Unit Acquired Weakness (Nervous system disorders) | 1 (1) | 1 (1)
Intercranial Pressure Increased (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Toxic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 1 (1)
Libido Decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Acute Renal Injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast Mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital Lesion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Embolism Venous (Vascular disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The AP-017 study was prematurely terminated by the sponsor after an interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT04839965/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/65/NCT04839965/SAP_001.pdf